CLINICAL TRIAL: NCT07102511
Title: Randomized, Placebo-Controlled, Double-Blind, Phase 3b Study to Evaluate the Efficacy and Safety of Lerodalcibep in Children and Adolescents, 6 to 17 Years of Age, With Heterozygous Familial Hypercholesterolemia on Stable Diet and Oral Lipid-Lowering Therapy
Brief Title: Randomized, Placebo-Controlled, Double-Blind, Phase 3b Study to Evaluate the Efficacy and Safety of Lerodalcibep in Children 6 to 17 Years, With Heterozygous FH
Acronym: LIBerate Kids
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-008
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Familial Hypercholesterolemia - Heterozygous
Keywords: inherited high cholesterol; high cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study drud administered by unblinded study staff memeber with no other role or contact with patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: lerodalcibep 300 mg (Active Comparator): monthly Subcutaneous injection
  Interventions: Biological: lerodalcibep 300 mg Monthly SC
- Arm 2: Placebo (Placebo Comparator): monthly subcutaneous injection
  Interventions: Biological: lerodalcibep 300 mg Monthly SC

INTERVENTIONS:
Biological: lerodalcibep 300 mg Monthly SC — lerodalcibep or placebo
  Other Names: placebo monthly SC

SUMMARY:
The goal of this clinical trial is to assess the LDL-Cholesterol reductions at Week 12 and Week 24 with monthly dosing of lerodalcibep (Lerochol) 300 mg administered subcutaneously by auto-injector (AI)/pre-filled pen (PFP) compared to placebo (dummy), in male and female pediatric patients 6 to 17 years of age, with inherited high cholesterol (HeFH) on a stable diet and maximally tolerated oral LDL C lowering drug therapy such as statins.

The main question[s] it aims to answer are:

How effective is Lerochol in reducing LDL cholesterol? How well is it tolerated and are there any safety concerns? Researchers will compare Lerochol to placebo (inert or dummy injection solution).

Participants will visit the clinic every month for months and be asked to fast overnight, but allowed to drink water, before clinic visits. Undergo physical exams, height and weight measurements, answer questions, have blood drawn from a vein in their arm, have blood pressure measurements, EKC heart tests, and receive monthly injections lasting about 5 seconds in their arms or abdomen with an autoinjector.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, Phase 3b study to evaluate the efficacy, safety, and tolerability of lerodalcibep 300 mg administered SC QM over a 24-week Treatment Period. Approximately 150 males and females, 6 to 17 years of age, with HeFH and who fulfill the inclusion and exclusion criteria will be enrolled at approximately 30 sites in the United States, Canada, Central and South America, Europe, South Africa, Asia, Australasia, and the Middle East. Patients will be randomized in a 2:1 ratio to lerodalcibep 300 mg (100 patients) or placebo (50 patients) administered SC QM. The study will consist of a Screening Period and a Treatment Period. The total study duration will be up to 35 weeks which includes up to an 11-week Screening Period (which may include up to an 8 week washout) and 24 weeks of study drug treatment

Following randomization and dosing on Day 1, patients will be seen in the clinic QM for 20 weeks and then at 2 week intervals for Weeks 22 and 24. All patients will receive doses of lerodalcibep 300 mg QM or placebo on Day 1 and Weeks 4, 8, 12, 16, and 20.

OBJECTIVES:

The co-primary objectives of this study are to assess the LDL-C reductions at Week 12 and Week 24 with monthly dosing of lerodalcibep 300 mg compared to placebo, in pediatric patients 6 to 17 years of age, with HeFH on a stable diet and maximally tolerated oral LDL C lowering drug therapy.

The secondary objectives of this study are the following:

* To assess the LDL-C-lowering effects of lerodalcibep with LDL-C calculated by Friedewald formula compared to placebo at Week 22 and the mean of Weeks 22 and 24;
* To assess the change in LDL-C, measured by preparative ultracentrifugation (PUC), from baseline (Week 0) with lerodalcibep compared to placebo at Week 24;
* To assess safety and tolerability of lerodalcibep in pediatric patients with HeFH;
* To assess the pharmacodynamic (PD) effects of 300 mg lerodalcibep QM on serum unbound (free) PCSK9 concentrations at Weeks 22 and 24;
* To assess the effects of lerodalcibep on serum lipids, including total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), non-HDL-C, very low-density lipoprotein cholesterol (VLDL-C), and triglycerides (TG);
* To assess the effects of lerodalcibep on ApoB and lipoprotein (a) (Lp[a]) serum concentrations compared to placebo at Weeks 12, 22, and 24, and the mean of Weeks 22 and 24;
* To assess the pharmacokinetics (PK) of lerodalcibep and total PCSK9 following 300 mg QM SC doses of lerodalcibep at Weeks 22 (peak post-dose) and 24 (trough post-dose); and
* To assess the frequency and level of anti-drug antibodies (ADAs) (immunogenicity) following multiple SC doses of lerodalcibep.

The exploratory objectives of this study are the following:

* To assess the LDL-C response based on underlying genetic variants associated with HeFH;
* To assess percentage of patients achieving current pediatric guidelines;
* To assess the effects on other lipid and cardiovascular risk biomarkers as appropriate;
* To assess the effects on physical development and endocrine tests as appropriate for age and sex; and
* To assess change from baseline in carotid intima-media thickness compared to placebo in children who do not tolerate statins, or have LDL-C levels >130 mg/dL despite >6 weeks, but <6 months, of statin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written and signed informed consent/assent prior to any study-specific procedure;
2. Male or female, 6 to 17 years of age (defined as from 6 to less than 18 years of age), at the first Screening Visit;
3. Weight of more than 18 kg (40 lbs) and BMI more than 17 and less than42 kg/m2;
4. Diagnosis of definite, probable, or possible HeFH based on clinical criteria (SB Register criteria or genotyping and at the defined eligibility visit (Screening Visit or post washout/stabilization); a calculated LDL-C (Friedewald) equal or above 130 mg/dL or, if the patient has additional risk factors as defined , a calculated LDL-C (Friedewald) equal or above100 mg/dL; and TG below 400 mg/dL while on stable lipid-lowering oral drug therapy (eg, maximally tolerated statin with or without ezetimibe); Note: Patients unable to tolerate approved doses of a statin may take lower than approved doses and less frequently than daily as long as the dose and dosing frequency is consistent per the Investigator's judgment. Patients with documented intolerance to statins may also participate;
5. On a stable diet and lipid-lowering oral therapies (statins, ezetimibe, bile-acid sequestrants) or combinations thereof for at least 6 weeks (excluded oral lipid-lowering agents include mipomersen, lomitapide, and gemfibrozil);
6. Patients on a PCSK9 mAb must undergo a washout period of >8 weeks after the last dose. For patients who have received an siRNA PCSK9 inhibitor the washout period is 360 days post last dose;
7. Females of childbearing potential must be using a highly effective form of contraception if sexually active and have negative urine pregnancy test at the last Screening Visit; Note: Highly effective methods of birth control include refraining from heterosexual sexual intercourse during the entire period of risk, birth control pills or patches, intrauterine devices (IUDs), sexual activity with a male partner who has had a vasectomy, condom or diaphragm or cervical cap with spermicide or IUD, oral, implantable, or injectable contraceptives.
8. Male patients will either be surgically sterile or agree to use the following forms of contraception: male or female condom with spermicide and a female partner who is sterile or who agrees to use the following contraceptives: diaphragm or cervical cap with spermicide; or IUD, oral, implantable, or injectable contraceptives; and
9. Male patients must refrain from sperm donation until 90 days following the last dose of study drug.

Exclusion Criteria:

1. Use of prohibited oral lipid-lowering agents mipomersen or lomitapide within 6 months of screening or gemfibrozil within 6 weeks of the Screening Visit;
2. LDL or plasma apheresis within 2 months prior to Day 1;
3. Documented history of HoFH defined as clinical and/or genetic with true HoFH (ie, identical pathogenic variants), compound heterozygous (ie, 2 different pathogenic LDLR variants) or combined heterozygous (2 different pathogenic FH variants such as LDLR plus ApoB or LDLR plus PCSK9 gain-of function);
4. History of any prior or active clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator, including but not limited to clinically significant pulmonary, hematologic, gastrointestinal, endocrine (excluding diabetes), immunologic, dermatologic, neurologic, or psychiatric disease, which in the Investigator's opinion, would not be suitable for the study from a patient safety consideration or could interfere with the results of the study;
5. Females of childbearing potential who are sexually active, not using or unwilling to use a highly effective form of contraception, pregnant or breastfeeding, or who have a positive urine pregnancy test at the last Screening Visit; Note: Highly effective methods of birth control include refraining from heterosexual sexual intercourse during the entire period of risk, birth control pills or patches, IUDs, sexual activity with a male partner who has had a vasectomy, condom or diaphragm or cervical cap with spermicide or IUD, oral, implantable, or injectable contraceptives.
6. Moderate to severe renal dysfunction, defined as an estimated glomerular filtration rate <30 mL/min/1.73m2 at the Screening Visit;
7. Active liver disease or hepatic dysfunction (eg, cirrhosis, alcoholic liver disease, known hepatitis B or hepatitis C, autoimmune hepatitis, liver failure, liver cancer), history of liver transplant, and/or AST or ALT >2.5 × the ULN based on age as determined by central laboratory analysis at screening (tests that result in ALT or AST up to 3 × ULN may have 1 repeat test to confirm eligibility during the Screening Period);
8. Uncontrolled thyroid disease: hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) below the lower limit of normal (LLN) or >1.5 × ULN, respectively, at the Screening Visit. If TSH is above/below these cut-off points, the patient can enter if the free triiodothyronine (FT3) is within the reference range. If controlled, then treatment should be stable for at least 3 months prior to the Screening Visit;
9. Uncontrolled Type 1 or Type 2 diabetes mellitus (defined as fasting glucose above 200 mg/dL and HbA1c of above 9%);
10. Uncontrolled serious cardiac arrhythmia (sustained ventricular tachycardia, frequent non sustained ventricular tachycardia, any ventricular fibrillation episode, wide-complex tachycardia, atrial fibrillation with rapid ventricular response, and severe second-degree or third degree atrioventricular block), myocardial infarction (MI), unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, placement of implantable cardioverter defibrillator or biventricular pacemaker, aortic valve surgery, or stroke within 3 months prior to enrollment (the day patient signs the informed consent/assent and first procedure is performed);
11. Planned cardiac surgery or revascularization;
12. New York Heart Association III-IV heart failure; or patients with last documented left ventricular ejection fraction <30% by standard of care assessments (eg, echocardiography, cardiac magnetic resonance imaging, nuclear imaging, computed tomography angiography, or angiography with ventriculogram), within 12 months;
13. Uncontrolled hypertension defined as a reproducible (ie, repeated 5 minutes apart) sitting blood pressure above 160 mmHg systolic or above 100 mmHg diastolic;
14. Enrolled in another investigational device or drug study, or less than 30 days or 5 half-lives since ending another investigational device or drug study(ies), or receiving other investigational agent(s); such as PCSK9 or ANGPTL3 or Lp(a) siRNA or locked nucleic acid reducing agents within 12 months of the Screening Visit;
15. Unexplained CK >5 × ULN, unless related to exercise or unusual activity in which case 1 repeat test is allowed;
16. Patients who cannot be available for Protocol-required study visits or procedures, to the best of the patient's and Investigator's knowledge;
17. A history, within 6 months prior to screening, of prescription drug abuse, illicit drug use, or alcohol abuse according to medical history;
18. Donated or lost a significant volume (>500 mL) of blood or plasma within 30 days prior to Day 1;
19. Had a blood transfusion within 4 weeks of randomization or known diagnosis of human immunodeficiency virus;
20. Previous treatment with lerodalcibep or any adnectin product;
21. Have any other finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study; or
22. An employee or family member of the Investigator or study site personnel.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male and female
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Low Density Lipoprotein cholesterol at week 12 | Week 12
  Change in LDL-C at week 12 relative to that of placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Kallend, MB BS, Study Director — Chief Medical Officer, LIB Therapeutics, LLC
Locations (3):
- Metabolic & Atherosclerosis Research Center, Cincinnati, Ohio, United States
- Lipid Clinic Wits University, Johannesburg, Gauteng, South Africa
- Ege Universitesi Tip Fakultesi, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No